CLINICAL TRIAL: NCT05570370
Title: Brain Oscillations, Sleep, and Arousal in Human Cognition - COL
Brief Title: Eardream Data Collection in Colombia Supported by ADDF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ADDF_COL
Record Dates: First submitted 2022-05-11; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADAD family members, mutation carriers: asymptomatic and presymptomatic individuals
  Interventions: Other: This is an observational study
- ADAD family members, non-mutation carriers: age-matched family members (non-mutation carriers) relative to the asymptomatic/presymptomatic group
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
Data collection based on this study will allow us to collect neurophysiological and cognitive data collected from in-ear EEG recordings of the Autosomal dominant alzheimer's disease population in Colombia

DETAILED DESCRIPTION:
There is solid neurophysiological evidence indicating that abnormal brain rhythms during sleep and noradrenergic dysfunction are core components of cognitive decline and AD onset, and their related pathophysiology. Crucially, irregularities in these neurophysiological mechanisms appear to occur in an asymptomatic and pre-symptomatic stage, but their potential to identify susceptibility for triggering neurodegeneration has yet to be established.

Thus, the possibility to identify such risk biomarkers in humans will require the acquisition of large-scale data related direct or indirect measurements of these physiological signatures. A possible key source to obtain such large-scale data related to sleep and noradrenergic function is the assessment of electroencephalographic recordings through non-obtrusive, low-cost, and reliable wearable sensors, alongside the use of advanced neuro-computational algorithms that link brain function and behavioral outcomes of LC function via pupilometry measurements.

ELIGIBILITY:
Participants fulfilling all of the following inclusion criteria are eligible for the study:

Informed Consent as documented by signature mutation and non-mutation carriers of ADAD populations Patients diagnosed with MCI and AD

Diseases or lesions of the nervous system (acute or residual included neurological and psychiatric diseases, except for MCI and AD in the patient population) Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.) Sleep disorders, known or suspected (e.g. Insomnia, sleep apnoea, restless leg syndrome, narcolepsy, etc.) mini mental state examination (MMSE) score > 24)

Participants are not eligible if they fulfill the following exclusion criteria:

Participation in another study with investigational drug/therapy/interventions within the 30 days preceding and during the present study (start date adapted accordingly) Suspected drug- or medication abuse, or on-label sleep medication use during the time of the study Infection/disease of the auditory canal or ear drum that could worsen with EAR-DREAM application, or allergies to in-Ear electrode materials (e.g., silver) Pregnancy (not safety related, but relevant for data interpretation procedures given that pregnancy can result in sleep patterns that are different from the baseline measurements we intend to characterize) Additional non-medical exclusion criteria may be defined for certain cognitive tasks (e.g. no glasses during experiments involving pupillometry).

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mutation and non-mutation carriers of ADAD populations Patients diagnosed with MCI and AD
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Density of slow-wave activity (SWA) readout from in-ear EEG recordings | Up to 7 nights of at-home recordings
  in-ear EEG will be monitored during 7 nights, the aggregated density of SWA over the 7 nights will be compared in both groups (mutation vs non-mutation carrier)
Relative phasic pupilometry responses in exploration vs exploration states in the cognitive task | experimental session at day 1
  atent variables of the LC-noradrenergic neuro-computational model based on our cognitive task will indicate the state in wich the participant is (exploration vs exploitation). The relative phasic pupilometry responses in these two states will serve as a proxy of the degree of LC-noradrenergic reaction to these states. The relative reactivity will be compared in both groups (mutation vs non-mutation carriers)

SECONDARY OUTCOMES:
Relative time-frequency decomposition responses in exploration vs exploration states in the cognitive task measured with EEG | experimental session at day 1
  We will evaluate the the differences spatio-temporal changes in the power spectrum depending on the state in wich the participant is (exploration vs exploitation) in the cognitive task. The relative changes will be compared in both groups (mutation vs non-mutation carriers)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Universitaria de Antioquia, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: Undecided